CLINICAL TRIAL: NCT03768531
Title: Safety and Tolerability Study of Combination Nivolumab and Cabiralizumab as Neoadjuvant and Adjuvant Therapy for Resectable Biliary Tract Cancer
Brief Title: Safety and Tolerability Study of Nivolumab and Cabiralizumab for Resectable Biliary Tract Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects were enrolled
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J18162; IRB00185328 (Other: JHM IRB)
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Resectable Biliary Tract Cancer
Keywords: Nivolumab; Cabiralizumab; Immunotherapy; Anti-PD-1; Anti-CSF-1R; Biliary tract cancers (BTC); Neoadjuvant chemotherapy; Adjuvant chemotherapy; Tumor microenvironment
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Nivolumab (Experimental)
  Interventions: Drug: Nivolumab
- Arm B: Nivolumab and Cabrilizumab (Experimental): Nivolumab 3 mg/kg will be given intravenously (IV) through a vein in the arm over 30 minutes, a 30 minute rest, followed by cabiralizumab every 2 weeks. (Cycle length 2 weeks).
  Interventions: Drug: Nivolumab; Drug: Cabrilizumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3 mg/kg will be given intravenously (IV) through a vein in the arm over 30 minutes every 2 weeks. (Cycle length 2 weeks).
  Other Names: OPDIVO; BMS-936558-01
Drug: Cabrilizumab — Cabiralizumab 4 mg/kg given IV for 30 minutes, 30 minutes after Nivolumab infusion is completed, every 2 weeks. (Cycle length 2 weeks).
  Other Names: FPA008, BMS-986227
  Arms: Arm B: Nivolumab and Cabrilizumab

SUMMARY:
The purposed of this research is to study the safety and clinical activity of the combination of nivolumab and cabiralizumab in people with resectable biliary tract cancers (BTC).

ELIGIBILITY:
Inclusion Criteria:

* Has confirmed biliary tract cancer
* Ability to understand and willingness to sign a written informed consent document.
* Age ≥18 years
* Have biopsiable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patient must have adequate organ function defined by the study-specified laboratory tests.
* Must use acceptable form of birth control while on study.

Exclusion Criteria:

* Has active autoimmune disease that requires systemic treatment.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years or that is expected to require active treatment within two years.
* Prior treatment with immunotherapy agents (including, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4, etc.).
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has evidence of an uncontrolled, active infection requiring parenteral anti-bacterial, anti-viral or anti-fungal therapy ≤ 7 days prior to administration of study medication.
* Has received a blood transfusion within 72 hours prior to first dose of study drug administration
* Unwilling or unable to follow the study schedule for any reason.
* Major surgery within 4 weeks prior to initiation of study treatment.
* Patient with uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant muscle disorders or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women.
* Have known history of infection with HIV, hepatitis B, or hepatitis C.
* Received any prophylactic vaccine within 30 days of first dose of study drug treatment.
* Has a history of allergy to study treatments or any of its components of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing study drug-related toxicities | 4 years
  Number of participants experiencing drug-related adverse events as defined by CTCAE v5.0

SECONDARY OUTCOMES:
Overall survival (OS) | 4 years
  Number of months from the date of first treatment until death or end of follow-up.
Disease free survival (DFS) | up to 4 years
  Number of months until disease recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Murphy, MD, Principal Investigator — Johns Hopkins Medical Institution

IPD SHARING:
Plan to Share IPD: No